CLINICAL TRIAL: NCT06549465
Title: A Phase 2, Open-label Study Evaluating Dosimetry, Randomized Dose Optimization, Dose Escalation and Efficacy of Ac-225 Rosopatamab Tetraxetan in Participants With PSMA PET-Positive Castration-Resistant Prostate Cancer
Brief Title: Study Evaluating Dosimetry, Randomized Dose Optimization, Dose Escalation and Efficacy of Ac-225 Rosopatamab Tetraxetan in Participants With PSMA PET-Positive Castration-Resistant Prostate Cancer (CRPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Convergent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CONVERGE-01
Record Dates: First submitted 2024-07-31; First posted 2024-08-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: PSMA PET-Positive Castration-Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: 148 ± 37 MBq In-111 rosopatamab tetraxetan (Experimental)
  Interventions: Biological: In-111 rosopatamab tetraxetan
- Part 2: 45 kBq/kg Ac-225 rosopatamab tetraxetan (Experimental)
  Interventions: Biological: 45 kBq/kg Ac-225 rosopatamab tetraxetan
- Part 2: 60 kBq/kg Ac-225 rosopatamab tetraxetan (Experimental)
  Interventions: Biological: 60 kBq/kg Ac-225 rosopatamab tetraxetan
- Part 3: Dose Escalation and Expansion (Experimental): Participants previously treated with Lu-177-PSMA-radioligand therapy will be assigned to receive one of the three dose levels (45 kBq/kg, 55 kBq/kg, or 60 kBq/kg) depending on the dose limiting toxicities (DLTs) observed.
  Interventions: Biological: 45 kBq/kg Ac-225 rosopatamab tetraxetan; Biological: 55 kBq/kg Ac-225 rosopatamab tetraxetan; Biological: 60 kBq/kg Ac-225 rosopatamab tetraxetan

INTERVENTIONS:
Biological: In-111 rosopatamab tetraxetan — A single dose of 148 ± 37 MBq In-111 rosopatamab tetraxetan will be administered as an IV infusion over a period of 10 minutes.
  Arms: Part 1: 148 ± 37 MBq In-111 rosopatamab tetraxetan
Biological: 45 kBq/kg Ac-225 rosopatamab tetraxetan — 45 kBq/kg Ac-225 rosopatamab tetraxetan will be administered as an IV infusion over a period of 10 minutes. Doses will be given two weeks apart for a total of two doses.
  Arms: Part 2: 45 kBq/kg Ac-225 rosopatamab tetraxetan; Part 3: Dose Escalation and Expansion
Biological: 55 kBq/kg Ac-225 rosopatamab tetraxetan — 55 kBq/kg Ac-225 rosopatamab tetraxetan will be administered as an IV infusion over a period of 10 minutes. Doses will be given two weeks apart for a total of two doses.
  Arms: Part 3: Dose Escalation and Expansion
Biological: 60 kBq/kg Ac-225 rosopatamab tetraxetan — 60 kBq/kg Ac-225 rosopatamab tetraxetan will be administered as an IV infusion over a period of 10 minutes. Doses will be given two weeks apart for a total of two doses.
  Arms: Part 2: 60 kBq/kg Ac-225 rosopatamab tetraxetan; Part 3: Dose Escalation and Expansion

SUMMARY:
This is a three-part study evaluating the safety and efficacy of a PSMA-directed radioantibody (rosopatamab tetraxetan, conjugated to either In-111 or Ac-225). Part 1 will consist of one administration of In-111-rosopatamab tetraxetan to characterize the biodistribution of the radioantibody to target organs and prostate cancer lesions. Participants then will be enrolled into either Part 2 (Dose Optimization) or Part 3 (Dose Escalation and Expansion) depending on their prior treatment history. Participants qualifying for Part 2 will be randomized to receive Ac-225 rosopatamab tetraxetan in a single fractionated cycle (dose administration on Day 1 and Day 15) at either 45 or 60 kBq/Kg. Participants qualifying for Part 3 must have received prior Lu-177-PSMA-radioligand therapy and will receive Ac-225 rosopatamab tetraxetan in a single fractionated cycle at 45, 55, or 60 kBq/Kg. Dose limiting toxicities (DLTs) will be monitored in Part 3 to determine the recommended phase 2 dose (RP2D), and the study may enroll additional participants to be treated with the RP2D dose level. Participants enrolled into any part will attend study visits which will include blood samples, electrocardiogram (ECG), radiographic imaging, and physical examinations along with other assessments.

ELIGIBILITY:
Inclusion Criteria:

* Progressive CRPC defined as castrate levels of testosterone and progressing by at least one of the following criteria:

  1. Serum PSA progression consisting of two consecutive increases in PSA measured at least 1 week apart. The minimal study baseline value is 2.0 ng/mL
  2. Soft tissue progression defined as a ≥20% increase in the sum of the diameter (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest sum of the diameter since the previous treatment was started or the appearance of one or more new lesions by CT/magnetic resonance imaging (MRI)
  3. Progression of bone disease defined by PCWG3 as evaluable disease or new bone lesions by bone scan
  4. Identification of new soft tissue or bone lesions on PSMA PET imaging
* Metastatic disease defined as either or both of the following:

  1. Parts 1, 2 and 3: Documented M1 disease on conventional imaging (CT/MRI of the chest/abdomen/pelvis and/or Technetium 99m [99mTc] whole-body bone scan)
  2. Parts 1 and 2 only: Identification of bone lesion(s), extra-pelvic soft tissue lesion(s), or visceral metastases on PSMA PET imaging with an FDA-approved imaging agent
* PSMA PET-positive disease, defined as at least one PSMA-positive metastatic lesion and no PSMA-negative lesions
* Progression following treatment with ADT and at least one ARSI (e.g., enzalutamide, apalutamide, darolutamide, and/or abiraterone acetate)
* The standard of care use (in the setting of metastatic CRPC with significant burden of active bone metastases) of antiresorptive bone-targeted agents (e.g., zoledronic acid, denosumab) is required for all participants without a contraindication, for at least 4 weeks prior to study drug administration
* Participants with HIV are eligible if they are well-controlled (i.e, an undetectable HIV viral load (<50 copies/mL) within 6 months of enrollment and a stable ART regimen for at least 6 months prior to enrollment) and at low risk for HIV-related illness

Part 3 Only:

* Prior treatment with Lu-177-PSMA-radioligand therapy
* Prior treatment with up to only one taxane-based chemotherapy regimen is allowed

Exclusion Criteria:

* Superscans by nuclear medicine/99mTc bone scan
* A known malignancy that is progressing or has required active treatment within the past 3 years other than CRPC, which is expected to alter life expectancy or may interfere with CRPC disease assessment
* Prior platinum-based chemotherapy
* Prior PARP inhibitors (e.g., olaparib or rucaparib)
* Prior treatment with Radium-223, Actinium-225, Strontium-89, Samarium-153, Rheunium-186, or Rhenium-188
* Participants receiving anti-coagulants or anti-platelet drugs (e.g., aspirin or nonsteroidal anti-inflammatory drugs [NSAIDs]) who cannot discontinue use if platelet count decreases to <50,000

Part 2 Only:

* Prior chemotherapy for CRPC. Prior taxane chemotherapy for HSPC is allowed if discontinued ≥1 year prior to randomization
* Prior radiopharmaceutical therapy (e.g., Ra-223, Lu-177-PSMA-617, or Lu-177-PSMA-I&T)
* Prior PSMA-targeted therapy

Part 3 Only:

* Prior PSMA-targeted therapy (e.g., antibody-drug conjugates or CAR-T therapy), except for Lu-177-PSMA-radioligand therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Visual evaluation on whole body planar scans (days 1 and 4) with comparison to reference scans for the presence of radiolabeled rosopatamab textraxetan in organs of interest (e.g., liver, circulation, spleen) to determine biodistribution | Day 1 and Day 4
Part 2: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) overall, by severity, and leading to discontinuation of study intervention | Screening through Week 12
Part 2: Proportion of participants who achieve a greater than or equal to 50% decline in prostate-specific antigen (PSA50) | Through end of study (approximately 3 years) or until PSA progression as defined by PCWG3 criteria
Part 3: Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) overall, by severity, and leading to discontinuation of study intervention | Screening through Week 12
Part 3: Determine the recommended Phase 2 dose (RP2D) of Ac-225 rosopatamab tetraxetan | Day 1 through 6 weeks
Part 3 (Participants treated at RP2D): Proportion of participants who achieve a greater than or equal to 50% decline in prostate-specific antigen (PSA50) | Through end of study (approximately 3 years) or until PSA progression as defined by PCWG3 criteria

SECONDARY OUTCOMES:
Part 2: Determine the clearance of rosopatamab tetraxetan and Ac-225 rosopatamab tetraxetan via measurement of whole blood and serum levels at specified serial timepoints | Through Week 8
Part 2: Radioactivity levels of Ac-225 rosopatamab tetraxetan | Through Day 21
Part 2: Radiation dosimetry of Ac-225 rosopatamab tetraxetan: Absorbed radiation dose (expressed as Gy/MBq) in normal organs | Day 1 through Day 15
Part 2: Biochemical progression-free survival (bPFS) as assessed by the Prostate Cancer Working Group 3 (PCWG3) | Through end of study (approximately 3 years) or until disease progression
Part 3: Proportion of participants who achieve PSA50 | Through end of study (approximately 3 years)
Part 3: Determine the clearance of rosopatamab tetraxetan and Ac-225 rosopatamab tetraxetan from the circulation via measurement in the serum at specified serial timepoints | Through Week 8
Part 3: Radioactivity levels of Ac-225 rosopatamab tetraxetan | Through Week 8

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of California San Diego, San Diego, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - X Cancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Laura & Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian/Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No